CLINICAL TRIAL: NCT05545267
Title: Monitoring of Dialysis Vascular Accesses During Angioplasty Under Echodoppler (SAVE)
Brief Title: Monitoring of Dialysis Vascular Accesses During Angioplasty Under Echodoppler
Acronym: SAVE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier de Vichy (Other)
Responsible Party: Sponsor
Other Study IDs: SAVE1 - CHV 2018-2
Record Dates: First submitted 2022-09-07; First posted 2022-09-19 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Arteriovenous Fistula Stenosis
Keywords: blood vessel repair; arteriovenous fistula; ultrasound angioplasty
MeSH Terms: conditions — Arteriovenous Fistula | interventions — Angioplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Angioplasties — Transluminal angioplastie
  Other Names: Angioplasties performed under echo-doppler

SUMMARY:
Dialysis vascular accesses called arteriovenous fistulas ( AVF) are essential to ensure extra-renal purification by hemodialysis for patients with chronic end-stage renal disease. Complications of dialysis AVF cause significant morbidity and hospitalization. Dialysis AVF angioplasties are frequently used to treat stenosis, the 1st complication concerning them and which announces the complete thrombosis which may be the definitive loss of the AVF. Historically performed under X-ray, the progression in the quality of ultrasound scanners allows today to perform this procedure under echo-Doppler guidance and thus to avoid both radiation and the injection of iodinated contrast products and their complications. It is thus possible to preserve residual renal function, a situation with a better prognosis, or to help the maturation of the AVF without precipitating the patient towards dialysis. The procedure can then be less costly, requiring a much lighter infrastructure.

The complication rates of ultrasound angioplasty remain poorly known because only a few series have been published. In addition, the evolution of the echo-Doppler parameters of the AVF is unknown during angioplasty and it is difficult to know which are the most reliable to distinguish during the procedure a "good angioplasty gesture" from an incomplete angioplasty to be continued. The proposed study would provide initial insight into the question posed.

DETAILED DESCRIPTION:
This is an observational, retrospective study on data from routine care. All angioplasties concerning major patients, meeting the inclusion criteria and performed during the inclusion period will be taken into account. (For this purpose, a list of procedures performed at the Vichy Hospital will be established via the angioplasty procedure reports.

In order to establish the evolution of the echographic parameters over time, the echographic data will also be collected from each follow-up report corresponding to each procedure until the end of the follow-up. These reports correspond to the normal post-intervention control ultrasounds at 1 month, 3 months and the annual visits. If intermediate ultrasounds are available, their reports will also be used.

In the case of a patient having an emergency angioplasty, the data of the control ultrasound triggering the intervention will be used as pre-intervention data.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Patient undergoing whose fistula is treated by angioplasty under echo-doplerat the Vichy Hospital Center between 01/01/2015 and 31/12/2019

Exclusion Criteria:

* Patients who are minors,
* Patients with an AVF with a flow rate < 100 mL/min.
* Patients with acute or chronic, segmental or total occlusion of an AVF segment
* Patients with acute or chronic, segmental or total thrombosis of an AVF segment
* Patients whose main obstacle is located on the arterial side.
* Intervention that required the use of X-rays.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with end-stage renal disease treated by dialysis whose AVF angioplasties is performed under echo-doppler at the Vcihy Hospital Center
Sampling Method: Non-Probability Sample
Enrollment: 144 (Actual)
Dates: Start 2021-09-17 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2022-10-31 (Estimated)

PRIMARY OUTCOMES:
morbidity and mortality | during intervention
  The primary outcome measure to evaluate morbidity and mortality will be the number of acute complications that occurred during the procedure and by type of complication (wall hematoma, thrombosis, rupture, spasm, injection site hematoma, pseudoaneurysm, failure)

SECONDARY OUTCOMES:
Post-angioplasty permeability | 2 years
  Post-angioplasty primary permeability, and post-angioplasty primary assisted permeability and post-angioplasty secondary permeability over the entire follow-up period
Stenosis diameter | pre-intervention, immediately after the intervention, 1 month
  Variation of the stenosis diameter
Endoluminal reference diameter | pre-intervention, immediately after the intervention, 1 month
  Variation of the endoluminal diameter
Maximum systolic velocity (VSmax) | pre-intervention, immediately after the intervention, 1 month
  Variation of the maximum systolic velocity
Ratio of VSmax to upstream | pre-intervention, immediately after the intervention, 1 month
  Varation of Ratio of VSmax to upstream
End-diastolic velocity | pre-intervention, immediately after the intervention, 1 month
  Variation of end-diastolic velocity
Diameter of the anastomosis | pre-intervention, immediately after the intervention, 1 month
  Variation of anastomosis diameter
Brachial artery Maximum flow | pre-intervention, immediately after the intervention, 1 month
  Variation of brachial artery maximum flow
Brachial artery end-diastolic velocity (EDV) | pre-intervention, immediately after the intervention, 1 month
  Varaition of Brachial artery end-diastolic velocity
Brachial artery maximum systolic velocity | pre-intervention, immediately after the intervention, 1 month
  Variation of brachial artery maximum systolic velocity
Brachial artery Resistance Index | pre-intervention, immediately after the intervention, 1 month
  Variation of brachial artery Resistance Index

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice ABBADIE, Study Director — Centre hopsitalier de Vichy
Locations (1):
- Centre Hospitalier de Vichy (CHV), Vichy, France

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, ICF
Time Frame: Immediately following publication ending 5 years following arti
Access Criteria: Researchers who provide a methodologically sound proposal. Proposals should be directed to Fabrice.Abbadie@ch-vichy.fr